CLINICAL TRIAL: NCT02173158
Title: A Phase 3, Single-Arm, Open-Label, Multicenter Study to Evaluate the Efficacy and Safety of Lomitapide in Japanese Patients With Homozygous Familial Hypercholesterolemia (HoFH) on Concurrent Lipid-Lowering Therapy
Brief Title: Efficacy and Safety of Lomitapide in Japanese Patients With HoFH on Concurrent Lipid-Lowering Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEGR-733-030
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-02

CONDITIONS: Familial Hypercholesterolemia - Homozygous
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — BMS201038

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lomitapide (Experimental): Maximum tolerated dose of lomitapide (up to 60mg/day) in addition to existing lipid lowering therapy including plasmapheresis or lipid apheresis.
  Interventions: Drug: lomitapide

INTERVENTIONS:
Drug: lomitapide
  Other Names: Juxtapid, Lojuxta

SUMMARY:
Study to Evaluate the Efficacy and Safety of Lomitapide in Japanese Patients with Homozygous Familial Hypercholesterolemia (HoFH) on Concurrent Lipid-Lowering Therapy.

DETAILED DESCRIPTION:
This is a Phase 3, single-arm, open-label, multicenter clinical trial to evaluate both the efficacy and long-term safety of lomitapide in Japanese patients with HoFH receiving maximally-tolerated, stable lipid-lowering therapy. This study is comprised of a run-in period, a primary 26-week Efficacy Phase, and a 30-week Safety Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese male and female patients aged ≥ 18 years of age who are receiving maximally tolerated, stable, lipid-lowering therapy
2. Diagnosis of functional HoFH
3. Body weight ≥ 40 kg and < 136 kg
4. Negative pregnancy test at screening

Exclusion Criteria:

1. Uncontrolled hypertension
2. History of chronic renal insufficiency
3. History of biopsy proven cirrhosis or abnormal liver function tests (LFTs) at screening
4. Any major surgical procedure occurring < 3 months prior to the screening visit
5. Cardiac insufficiency
6. Previous organ transplantation
7. History of a non-skin malignancy within the previous 3 years
8. Patients who are not able to limit their alcohol intake
9. Participation in an investigational drug study within 6 weeks prior to the screening visit
10. Known significant gastrointestinal bowel disease
11. Nursing mothers
12. Serious or unstable medical or psychological conditions
13. Requirement for certain prohibited medications known to be potentially hepatotoxic
14. Use of strong or moderate inhibitors of CYP3A4
15. Use of simvastatin at doses >10 mg per day
16. Documented diagnosis of any liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04-02 (Actual); Primary Completion 2015-04-03 (Actual); Study Completion 2015-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariko Harada-Shiba, M.D., Ph.D., Principal Investigator — National Cerebral and Cardiovascular Center Research Institute
Locations (6):
- Japan (6):
  - Kurume-shi, Fukuoka
  - Kanazawa, Ishikawa-ken
  - Osakashi, Osaka
  - Suita-shi, Osaka
  - Tokorozawa, Saitama
  - Bunkyo-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Period: Efficacy Phase
Arm/Group | Lomitapide
Started | 9
Completed | 8
Not Completed | 1
Not completed — Adverse Event | 1
Period: Safety Phase
Arm/Group | Lomitapide
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in LDL-C
Description: Mean percent change from baseline
Time Frame: Baseline to Week 26
Population: Full analysis set for the efficacy phase, included all subjects who received study drug and had a baseline and at least one post-baseline assessment
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lomitapide
Number analyzed (Participants) | 9
Percent change | -42.2 (18.16)

2. Secondary Outcome: Change in Total Cholesterol
Description: Mean percent change from baseline
Time Frame: Baseline to Week 56
Population: Full analysis set for the safety phase included all subjects who received study drug during the safety phase and had at least one assessment during the safety phase
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lomitapide
Number analyzed (Participants) | 8
Percent change | -25.9 (18.57)

3. Secondary Outcome: Change in Apo B
Description: Mean percent change from baseline
Time Frame: Baseline to Week 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lomitapide
Number analyzed (Participants) | 8
Percent change | -41.4 (21.90)

4. Secondary Outcome: Change in Triglycerides
Description: Mean percent change from baseline
Time Frame: Baseline to Week 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lomitapide
Number analyzed (Participants) | 8
Percent change | -44.4 (12.70)

5. Secondary Outcome: Change in Non-HDL-C
Description: Mean percent change from baseline
Time Frame: Baseline to Week 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lomitapide
Number analyzed (Participants) | 8
Percent change | -34.6 (22.50)

6. Secondary Outcome: Change in VLDL-C
Description: Mean percent change from baseline
Time Frame: Baseline to Week 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lomitapide
Number analyzed (Participants) | 8
Percent change | -44.8 (12.05)

7. Secondary Outcome: Change in Lp(a)
Description: Mean percent change from baseline
Time Frame: Baseline to Week 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lomitapide
Number analyzed (Participants) | 8
Percent change | -27.2 (23.50)

8. Secondary Outcome: Change in HDL-C
Description: Mean percent change from baseline
Time Frame: Baseline to Week 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lomitapide
Number analyzed (Participants) | 8
Percent change | 5.9 (19.64)

9. Secondary Outcome: Change in Apo AI
Description: Mean percent change from baseline
Time Frame: Baseline to Week 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lomitapide
Number analyzed (Participants) | 8
Percent change | -2.8 (11.61)

10. Secondary Outcome: Change in LDL-C
Description: Mean percent change from baseline
Time Frame: Baseline to Week 56
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Lomitapide
Number analyzed (Participants) | 8
Percent change | -37.5 (24.21)

ADVERSE EVENTS:
Groups:
- Efficacy Phase: Baseline to Week 26
- Safety Phase: Week 26 to Week 56
Arm/Group | Efficacy Phase | Safety Phase
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/8
Other Adverse Events (participants affected / at risk) | 9/9 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Efficacy Phase (N=9) | Safety Phase (N=8)
Chest pain (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efficacy Phase (N=9) | Safety Phase (N=8)
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Nausea (Gastrointestinal disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Nasopharyngitis (Infections and infestations) | 4 | 3
Gastroenteritis (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 1
Periodontitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0
Chest pain (General disorders) | 0 | 1
Device breakage (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 0
Chemical burn of skin (Injury, poisoning and procedural complications) | 0 | 1
Heat stroke (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1
Liver function test abnormal (Investigations) | 3 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Mylagia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Described in site contract